CLINICAL TRIAL: NCT02549040
Title: A Rapid Pharmacokinetic Trial of the Bioavailability of Four MK-1439 Nano Formulations in Healthy Adults
Brief Title: Bioavailability of Doravirine (MK-1439) Experimental Nano Formulations in Healthy Adults (MK-1439-046)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1439-046; 2015-002702-36 (EudraCT Number); MK-1439-046 (Other: Merck Protocol Number)
Record Dates: First submitted 2015-09-11; First posted 2015-09-14 (Estimated); Results first posted 2019-02-22 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Human Immunodeficiency Virus-1 (HIV-1)
MeSH Terms: interventions — doravirine; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doravirine fixed sequence treatment (Experimental): After a minimum 10 hour overnight fast, participants received a single oral dose during each of 5 periods. During Period 1, participants received Treatment B: Doravirine Type 1 dose (150 mg tablet [40% drug loaded granule]). During Period 2, participants received Treatment A: Doravirine 100 mg film coated tablet. During Period 3, participants received Treatment C: Doravirine Type 2 dose (150 mg tablet [30% drug loaded granule]). During Period 4, participants received Treatment D: Doravirine Type 3 dose (150 mg tablet [50% drug loaded granule]. During Period 5, participants received Treatment E: Doravirine Type 4 dose (100 mg tablet [30% drug loaded granule]). Each period was separated by a 14 day washout.
  Interventions: Drug: Treatment A: Doravirine 100 mg film coated tablet; Drug: Treatment B: Doravirine 150 mg tablet (40% drug loaded granule); Drug: Treatment C: Doravirine 150 mg tablet (30% drug loaded granule); Drug: Treatment D: Doravirine 150 mg tablet (50% drug loaded granule); Drug: Treatment E: Doravirine 100 mg tablet (30% drug loaded granule)

INTERVENTIONS:
Drug: Treatment A: Doravirine 100 mg film coated tablet — Single doravirine 100 mg film coated tablet administered orally at the start of Period 2
  Other Names: MK-1439
Drug: Treatment B: Doravirine 150 mg tablet (40% drug loaded granule) — Single doravirine NF Type 1 dose (150 mg tablet [40% drug loaded granule]) administered orally at the start of Period 1
  Other Names: MK-1439
Drug: Treatment C: Doravirine 150 mg tablet (30% drug loaded granule) — Single doravirine NF Type 2 dose (150 mg tablet [30% drug loaded granule])administered orally at the start of Period 3
  Other Names: MK-1439
Drug: Treatment D: Doravirine 150 mg tablet (50% drug loaded granule) — Single doravirine NF Type 3 dose (150 mg tablet [50% drug loaded granule])administered orally at the start of Period 4
  Other Names: MK-1439
Drug: Treatment E: Doravirine 100 mg tablet (30% drug loaded granule) — Single doravirine NF Type 4 dose (100 mg tablet [30% drug loaded granule]) administered orally at the start of Period 5
  Other Names: MK-1439

SUMMARY:
This study aims to evaluate and compare the relative bioavailability of different doravirine (MK-1439) experimental nano formulations (NFs) with that of a doravirine film coated tablet.

ELIGIBILITY:
Inclusion Criteria:

* healthy participants
* have been a non-smoker and/or have not used nicotine or nicotine-containing products for at least approximately 3 months

Exclusion Criteria:

* is a pregnant or a nursing female
* has a history of stroke, chronic seizures or major neurological disorder
* has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* has a history of neoplastic disease (including leukemia, lymphoma, malignant melanoma), or myeloproliferative disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-09-21 (Actual); Primary Completion 2015-12-24 (Actual); Study Completion 2015-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-1439 Fixed Sequence Treatment: After a minimum 10 hour overnight fast, participants received a single oral dose during each of 5 periods. During Period 1, participants received Treatment B: MK-1439 Type 1 dose (150 mg tablet [40% drug loaded granule]). During Period 2, participants received Treatment A: MK-1439 100 mg film coated tablet. During Period 3, participants received Treatment C: MK-1439 Type 2 dose (150 mg tablet [30% drug loaded granule]). During Period 4, participants received Treatment D: MK-1439 Type 3 dose (150 mg tablet [50% drug loaded granule]. During Period 5, participants received Treatment E: MK-1439 Type 4 dose (100 mg tablet [30% drug loaded granule]). Each period was separated by a 14 day washout.
Period: Period 1
Arm/Group | MK-1439 Fixed Sequence Treatment
Started | 16
Completed | 16
Not Completed | 0
Period: Period 2
Arm/Group | MK-1439 Fixed Sequence Treatment
Started | 16
Completed | 16
Not Completed | 0
Period: Period 3
Arm/Group | MK-1439 Fixed Sequence Treatment
Started | 16
Completed | 16
Not Completed | 0
Period: Period 4
Arm/Group | MK-1439 Fixed Sequence Treatment
Started | 16
Completed | 16
Not Completed | 0
Period: Period 5
Arm/Group | MK-1439 Fixed Sequence Treatment
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MK-1439 Fixed Sequence Treatment
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC0-inf) of MK-1439 Following a Single Administration of MK-1439
Description: During each of the 5 treatment periods, blood samples were collected pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 12, 24, 48, and 72 hours post-dose to determine AUC0-inf after a single administration of MK-1439.
Time Frame: Periods 1 to 5 at the following time points: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 12, 24, 48, and 72 hours post-dose
Population: Participants who complied with the protocol sufficiently to ensure that the data exhibited the effects of treatment, according to the underlying scientific model. Participants were excluded from descriptive statistics for AUC0-inf if there were insufficient data in the terminal phase to characterize half-life (t1/2).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µM*h
Groups:
- Treatment B: MK-1439 150 mg Tablet (40% Drug Loaded Granule): Participants received a single MK-1439 Type 1 dose (150 mg tablet [40% drug loaded granule]) administered orally at the start of Period 1
- Treatment A: MK-1439 100 mg Film Coated Tablet: Participants received a single MK-1439 100 mg film coated tablet administered orally at the start of Period 2
- Treatment C: MK-1439 150 mg Tablet (30% Drug Loaded Granule): Participants received a single MK-1439 Type 2 dose (150 mg tablet [30% drug loaded granule]) administered orally at the start of Period 3
- Treatment D: MK-1439 150 mg Tablet (50% Drug Loaded Granule): Participants received a single MK-1439 Type 3 dose (150 mg tablet [50% drug loaded granule]) administered orally at the start of Period 4
- Treatment E: MK-1439 100 mg Tablet (30% Drug Loaded Granule): Participants received a single MK-1439 Type 4 dose (100 mg tablet [30% drug loaded granule]) administered orally at the start of Period 5
Arm/Group | Treatment B: MK-1439 150 mg Tablet (40% Drug Loaded Granule) | Treatment A: MK-1439 100 mg Film Coated Tablet | Treatment C: MK-1439 150 mg Tablet (30% Drug Loaded Granule) | Treatment D: MK-1439 150 mg Tablet (50% Drug Loaded Granule) | Treatment E: MK-1439 100 mg Tablet (30% Drug Loaded Granule)
Number analyzed (Participants) | 13 | 16 | 15 | 12 | 15
µM*h | 28.6 (34.6) | 31.9 (33.9) | 35.5 (29.6) | 29.1 (30.3) | 28.0 (27.5)
Statistical Analysis 1: Comparison: Treatment B: MK-1439 150 mg Tablet (40% Drug Loaded Granule) vs Treatment A: MK-1439 100 mg Film Coated Tablet; Comparison of Treatment B: MK-1439 150 mg tablet (40% drug loaded granule) vs. Treatment A: MK-1439 100 mg film coated tablet; Test type: Other; Geometric mean ratio = 0.96, 90% CI 2-sided [0.85 to 1.09]
Statistical Analysis 2: Comparison: Treatment A: MK-1439 100 mg Film Coated Tablet vs Treatment C: MK-1439 150 mg Tablet (30% Drug Loaded Granule); Comparison of Treatment C: MK-1439 150 mg tablet (30% drug loaded granule) vs. Treatment A: MK-1439 100 mg film coated tablet; Test type: Other; Geometric mean ratio = 1.13, 90% CI 2-sided [1.02 to 1.26]
Statistical Analysis 3: Comparison: Treatment A: MK-1439 100 mg Film Coated Tablet vs Treatment D: MK-1439 150 mg Tablet (50% Drug Loaded Granule); Comparison of Treatment D: MK-1439 150 mg tablet (50% drug loaded granule) vs. Treatment A: MK-1439 100 mg film coated tablet; Test type: Other; Geometric mean ratio = 0.99, 90% CI 2-sided [0.88 to 1.11]
Statistical Analysis 4: Comparison: Treatment A: MK-1439 100 mg Film Coated Tablet vs Treatment E: MK-1439 100 mg Tablet (30% Drug Loaded Granule); Comparison of Treatment E: MK-1439 100 mg tablet (30% drug loaded granule) vs. Treatment A: MK-1439 100 mg film coated tablet; Test type: Other; Geometric mean ratio = 0.89, 90% CI 2-sided [0.80 to 0.99]

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Last Time (AUC0-last) With Quantifiable MK-1439 Following a Single Administration of MK-1439
Description: During each of the 5 treatment periods, blood samples were collected pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 12, 24, 48, and 72 hours post-dose to determine AUC0-last after a single administration of MK-1439.
Time Frame: Periods 1 to 5 at the following time points: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 12, 24, 48, and 72 hours post-dose
Population: Participants who complied with the protocol sufficiently to ensure that the data exhibited the effects of treatment, according to the underlying scientific model.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM*h
Arm/Group | Treatment B: MK-1439 150 mg Tablet (40% Drug Loaded Granule) | Treatment A: MK-1439 100 mg Film Coated Tablet | Treatment C: MK-1439 150 mg Tablet (30% Drug Loaded Granule) | Treatment D: MK-1439 150 mg Tablet (50% Drug Loaded Granule) | Treatment E: MK-1439 100 mg Tablet (30% Drug Loaded Granule)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
μM*h | 26.3 (29.3) | 29.9 (31.1) | 32.7 (26.3) | 27.0 (28.4) | 26.3 (27.0)
Statistical Analysis 1: Comparison: Treatment B: MK-1439 150 mg Tablet (40% Drug Loaded Granule) vs Treatment A: MK-1439 100 mg Film Coated Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio = 0.88, 90% CI 2-sided [0.79 to 0.98]
Statistical Analysis 2: Comparison: Treatment A: MK-1439 100 mg Film Coated Tablet vs Treatment C: MK-1439 150 mg Tablet (30% Drug Loaded Granule); [analysis description as in outcome 1, analysis 2]; Test type: Other; Geometric mean ratio = 1.09, 90% CI 2-sided [0.98 to 1.21]
Statistical Analysis 3: Comparison: Treatment A: MK-1439 100 mg Film Coated Tablet vs Treatment D: MK-1439 150 mg Tablet (50% Drug Loaded Granule); [analysis description as in outcome 1, analysis 3]; Test type: Other; Geometric mean ratio = 0.90, 90% CI 2-sided [0.81 to 1.00]
Statistical Analysis 4: Comparison: Treatment A: MK-1439 100 mg Film Coated Tablet vs Treatment E: MK-1439 100 mg Tablet (30% Drug Loaded Granule); [analysis description as in outcome 1, analysis 4]; Test type: Other; Geometric mean ratio = 0.88, 90% CI 2-sided [0.79 to 0.97]

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of MK-1439 Following a Single Administration of MK-1439
Description: During each of the 5 treatment periods, blood samples were collected pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose to determine Cmax after a single administration of MK-1439.
Time Frame: Periods 1 to 5 at the following time points: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Treatment B: MK-1439 150 mg Tablet (40% Drug Loaded Granule) | Treatment A: MK-1439 100 mg Film Coated Tablet | Treatment C: MK-1439 150 mg Tablet (30% Drug Loaded Granule) | Treatment D: MK-1439 150 mg Tablet (50% Drug Loaded Granule) | Treatment E: MK-1439 100 mg Tablet (30% Drug Loaded Granule)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
nM | 1070 (26.5) | 1520 (32.5) | 1320 (27.8) | 1060 (27.0) | 1160 (24.2)
Statistical Analysis 1: Comparison: Treatment B: MK-1439 150 mg Tablet (40% Drug Loaded Granule) vs Treatment A: MK-1439 100 mg Film Coated Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio = 0.70, 90% CI 2-sided [0.61 to 0.82]
Statistical Analysis 2: Comparison: Treatment A: MK-1439 100 mg Film Coated Tablet vs Treatment C: MK-1439 150 mg Tablet (30% Drug Loaded Granule); [analysis description as in outcome 1, analysis 2]; Test type: Other; Geometric mean ratio = 0.87, 90% CI 2-sided [0.75 to 1.01]
Statistical Analysis 3: Comparison: Treatment A: MK-1439 100 mg Film Coated Tablet vs Treatment D: MK-1439 150 mg Tablet (50% Drug Loaded Granule); [analysis description as in outcome 1, analysis 3]; Test type: Other; Geometric mean ratio = 0.70, 90% CI 2-sided [0.60 to 0.81]
Statistical Analysis 4: Comparison: Treatment A: MK-1439 100 mg Film Coated Tablet vs Treatment E: MK-1439 100 mg Tablet (30% Drug Loaded Granule); [analysis description as in outcome 1, analysis 4]; Test type: Other; Geometric mean ratio = 0.76, 90% CI 2-sided [0.66 to 0.86]

4. Primary Outcome: Plasma Concentration of MK-1439 at 24 Hours Post-dose (C24hr) Following a Single Administration of MK-1439
Description: During each of the 5 treatment periods, blood samples were collected 24 hours after dosing to determine C24hr after a single administration of MK-1439.
Time Frame: Periods 1 to 5: 24 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Treatment B: MK-1439 150 mg Tablet (40% Drug Loaded Granule) | Treatment A: MK-1439 100 mg Film Coated Tablet | Treatment C: MK-1439 150 mg Tablet (30% Drug Loaded Granule) | Treatment D: MK-1439 150 mg Tablet (50% Drug Loaded Granule) | Treatment E: MK-1439 100 mg Tablet (30% Drug Loaded Granule)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
nM | 395 (31.9) | 483 (33.3) | 508 (23.2) | 412 (28.0) | 402 (32.0)
Statistical Analysis 1: Comparison: Treatment B: MK-1439 150 mg Tablet (40% Drug Loaded Granule) vs Treatment A: MK-1439 100 mg Film Coated Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio = 0.82, 90% CI 2-sided [0.72 to 0.93]
Statistical Analysis 2: Comparison: Treatment A: MK-1439 100 mg Film Coated Tablet vs Treatment C: MK-1439 150 mg Tablet (30% Drug Loaded Granule); [analysis description as in outcome 1, analysis 2]; Test type: Other; Geometric mean ratio = 1.05, 90% CI 2-sided [0.94 to 1.18]
Statistical Analysis 3: Comparison: Treatment A: MK-1439 100 mg Film Coated Tablet vs Treatment D: MK-1439 150 mg Tablet (50% Drug Loaded Granule); [analysis description as in outcome 1, analysis 3]; Test type: Other; Geometric mean ratio = 0.85, 90% CI 2-sided [0.76 to 0.96]
Statistical Analysis 4: Comparison: Treatment A: MK-1439 100 mg Film Coated Tablet vs Treatment E: MK-1439 100 mg Tablet (30% Drug Loaded Granule); [analysis description as in outcome 1, analysis 4]; Test type: Other; Geometric mean ratio = 0.83, 90% CI 2-sided [0.74 to 0.94]

5. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event
Description: An adverse event is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not it is considered related to the study drug.
Time Frame: Up to 16 days after last dose of study treatment (up to approximately 92 days)
Population: All participants who received at least 1 administration of the trial drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment B: MK-1439 150 mg Tablet (40% Drug Loaded Granule) | Treatment A: MK-1439 100 mg Film Coated Tablet | Treatment C: MK-1439 150 mg Tablet (30% Drug Loaded Granule) | Treatment D: MK-1439 150 mg Tablet (50% Drug Loaded Granule) | Treatment E: MK-1439 100 mg Tablet (30% Drug Loaded Granule)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Participants | 2 | 5 | 4 | 6 | 1

6. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event
Description: as for outcome 5
Time Frame: Up to 4 days after last dose of study treatment (up to approximately 76 days)
Population: All participants who received at least 1 administration of the trial drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment B: MK-1439 150 mg Tablet (40% Drug Loaded Granule) | Treatment A: MK-1439 100 mg Film Coated Tablet | Treatment C: MK-1439 150 mg Tablet (30% Drug Loaded Granule) | Treatment D: MK-1439 150 mg Tablet (50% Drug Loaded Granule) | Treatment E: MK-1439 100 mg Tablet (30% Drug Loaded Granule)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Participants | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to 48 Hours (AUC0-48 hr) Post-dose of MK-1439 Following a Single Administration of MK-1439
Description: During each of the 5 treatment periods, blood samples were collected pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 12, 24, 48 hours after dosing to determine AUC0-48hr after a single administration of MK-1439.
Time Frame: Periods 1 to 5 at the following time points: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 12, 24, and 48 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µM*h
Arm/Group | Treatment B: MK-1439 150 mg Tablet (40% Drug Loaded Granule) | Treatment A: MK-1439 100 mg Film Coated Tablet | Treatment C: MK-1439 150 mg Tablet (30% Drug Loaded Granule) | Treatment D: MK-1439 150 mg Tablet (50% Drug Loaded Granule) | Treatment E: MK-1439 100 mg Tablet (30% Drug Loaded Granule)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
µM*h | 22.8 (27.5) | 27.2 (29.2) | 28.8 (24.8) | 23.2 (27.3) | 23.3 (25.9)
Statistical Analysis 1: Comparison: Treatment B: MK-1439 150 mg Tablet (40% Drug Loaded Granule) vs Treatment A: MK-1439 100 mg Film Coated Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio = 0.84, 90% CI 2-sided [0.75 to 0.94]
Statistical Analysis 2: Comparison: Treatment A: MK-1439 100 mg Film Coated Tablet vs Treatment C: MK-1439 150 mg Tablet (30% Drug Loaded Granule); [analysis description as in outcome 1, analysis 2]; Test type: Other; Geometric mean ratio = 1.06, 90% CI 2-sided [0.95 to 1.18]
Statistical Analysis 3: Comparison: Treatment A: MK-1439 100 mg Film Coated Tablet vs Treatment D: MK-1439 150 mg Tablet (50% Drug Loaded Granule); [analysis description as in outcome 1, analysis 3]; Test type: Other; Geometric mean ratio = 0.85, 90% CI 2-sided [0.76 to 0.95]
Statistical Analysis 4: Comparison: Treatment A: MK-1439 100 mg Film Coated Tablet vs Treatment E: MK-1439 100 mg Tablet (30% Drug Loaded Granule); [analysis description as in outcome 1, analysis 4]; Test type: Other; Geometric mean ratio = 0.86, 90% CI 2-sided [0.77 to 0.96]

ADVERSE EVENTS:
Time Frame: Up to 16 days following the last dose of study treatment (up to approximately 92 days)
Arm/Group | Treatment B: MK-1439 150 mg Tablet (40% Drug Loaded Granule) | Treatment A: MK-1439 100 mg Film Coated Tablet | Treatment C: MK-1439 150 mg Tablet (30% Drug Loaded Granule) | Treatment D: MK-1439 150 mg Tablet (50% Drug Loaded Granule) | Treatment E: MK-1439 100 mg Tablet (30% Drug Loaded Granule)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 2/16 | 5/16 | 4/16 | 6/16 | 1/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment B: MK-1439 150 mg Tablet (40% Drug Loaded Granule) (N=16) | Treatment A: MK-1439 100 mg Film Coated Tablet (N=16) | Treatment C: MK-1439 150 mg Tablet (30% Drug Loaded Granule) (N=16) | Treatment D: MK-1439 150 mg Tablet (50% Drug Loaded Granule) (N=16) | Treatment E: MK-1439 100 mg Tablet (30% Drug Loaded Granule) (N=16)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling of body temperture change (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 3 (4) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menstrual discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.